CLINICAL TRIAL: NCT01084226
Title: Dietary Intervention Trial of Alkylresorcinols and Plant Sterols in High-Fibre Rye Bread and Their Effects on Serum Lipids in Normo- and Mildly Hypercholesterolemic Subjects
Brief Title: Rye Bread Trial; Antioxidative and Cholesterol Lowering Effects
Acronym: Rye-2008
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Samfundet Folkhälsan (Unknown); Sigrid Jusélius Foundation (Other); Fazer (Other)
Model: Parallel | Masking: Triple
Other Study IDs: 1/13/03/00/08
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Hypercholesterol
Keywords: Rye fiber; Alkylresorcinols; Plant sterols; Cholesterol; Antioxidant; Effects of plant sterols in rye bread on serum lipids; Effects of alkylresorcinols in rye fiber on LDL particles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Sterol (Active Comparator): Additional plant sterols incorporated in the rye bread
  Interventions: Dietary Supplement: Rye-2008
- control (Placebo Comparator): No added plant sterol in the identical-looking rye bread
  Interventions: Dietary Supplement: Rye-2008

INTERVENTIONS:
Dietary Supplement: Rye-2008

SUMMARY:
The purpose of this study is to investigate the antioxidative effects of alkylresorcinols (AR), originating from the rye fiber, on serum LDL particles and the use of AR or it's metabolites as biomarkers for rye fiber intake and the effect of additional plants sterols, incorporated in the rye bread, on serum total and LDL cholesterol concentration.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* volunteer
* hemoglobin above 125 mmol/L in females, above 135 mmol/L in males

Exclusion Criteria:

* taking drugs affecting plasma lipids or gastrointestinal track
* severe illness
* use of antibiotics within 3 months before entering the study
* use of vitamin pills or fish oil 1 month before entering the study
* pregnancy or lactating

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2010-02

CONTACTS AND LOCATIONS:
Overall Officials: Matti J Tikkanen, M.D.. Prof., Study Director — Department of Medicine, University of Helsinki, Helsinki, Finland
Locations (1):
- Folkhälsan Research Center, Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Soderholm PP, Alfthan G, Tikkanen MJ, Adlercreutz H. Rye bread intake improves oxidation resistance of LDL in healthy humans. Atherosclerosis. 2012 Apr;221(2):583-6. doi: 10.1016/j.atherosclerosis.2012.01.030. Epub 2012 Jan 25. PMID 22336172
- [Derived] Soderholm PP, Alfthan G, Koskela AH, Adlercreutz H, Tikkanen MJ. The effect of high-fiber rye bread enriched with nonesterified plant sterols on major serum lipids and apolipoproteins in normocholesterolemic individuals. Nutr Metab Cardiovasc Dis. 2012 Jul;22(7):575-82. doi: 10.1016/j.numecd.2010.09.011. Epub 2011 Jan 6. PMID 21215605